CLINICAL TRIAL: NCT06061458
Title: Assessment of Children With Variable Hearing Amplification Devices by Speech Auditory Brainstem Response
Brief Title: Assessment of Children by Speech ABR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, kholoud omar, MD, Principle Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACDS
Record Dates: First submitted 2023-09-14; First posted 2023-09-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hearing Impaired Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): normal hearing
- the group with hearing aids (Experimental): children with hearing aids
  Interventions: Diagnostic Test: speech auditory brainstem response
- the group with cochlear implant (Experimental): children with cochlear implant
  Interventions: Diagnostic Test: speech auditory brainstem response
- the group with bimodal hearing (Experimental): children with bimodal hearing
  Interventions: Diagnostic Test: speech auditory brainstem response

INTERVENTIONS:
Diagnostic Test: speech auditory brainstem response — A diagnostic objective test to evaluate the speech process in hearing impaired children
  Arms: the group with bimodal hearing; the group with cochlear implant; the group with hearing aids

SUMMARY:
Assessment of children by speech auditory brainstem response which is an objective method to study the speech development

DETAILED DESCRIPTION:
Hearing loss in children can result in cognitive deficits in the central areas which are dependent upon hearing, therefore responsible for delay in speech development, poor language skills and disorders in psychological and mental behavior. It will also cause a decrease of the intellectual ability and socio-economic position of the child.

In children aged 3.5 years and older, pure tone audiometry is performed to determine the exact frequency-specific hearing threshold.

To obtain the auditory threshold in younger children, Skoe and Kraus reported that the auditory brainstem response has proven to be a clinically useful tool for assessing neural function at the brainstem level and is most commonly elicited by clicks or tone-bursts.

However, recent research has established that complex stimuli can also elicit the response such as Music, complex tones, and speech stimuli . A speech stimulus is particularly useful, as it can provide clues as to how temporal and spectral features are preserved in the brainstem.

The human soundscape is characterized by complex sounds with rich harmonic structure, dynamic amplitude modulations and rapid spectro-temporal fluctuations. This complexity is represented by temporal and spectral neural code within the auditory brainstem, two broad classes of time-locked responses can be defined namely transient and sustained responses .

Although complex sounds consist of both sustained and transient features, the response to a complex sound is not necessarily predictable from the response to click auditory brainstem response . For these reason, further studies had gradually transitioned to using sounds as stimuli as they are more complex .

The click auditory brainstem response is a clinical tool to assess the neural functionality of the auditory brainstem. The use of verbal stimuli in auditory brainstem response protocols has provided important information of how the speech stimuli are processed by the brainstem structure .

The perception of speech sounds seems to begin in the brainstem, which has an important role in the reading process and the phonological acquisition . Speech auditory brainstem response assessment allows the identification of fine-grained auditory processing deficits associated with real world communication which do not appear in click evoked auditory brainstem response .

The verbal stimulus most widely used in speech auditory brainstem response is a syllable composed of a consonant and a vowel , usually the syllables da. The verbal assessment provides information about how the speech syllable is encoded by auditory system. The trace of the speech auditory brainstem response can be identified in two parts:

The onset and the frequency following response . The first part represents the consonant and the second part represents the vowel .

So speech auditory brainstem response can be used as an objective measure of the hearing function, one of the great advantages of this method is that it is not influenced by environmental issues, which can disrupt the behavioral assessments . Even the best behavioral tests can be affected by multiple factors such as attention, motivation and alertness or fatigue .

Moreover, altered responses of speech auditory brainstem response may be associated with impaired speech perception specially in noise. These changes can cause a negative impact on communication and serious consequences for academic success in children. complex auditory brainstem response can also help to identify those individuals who are most likely to benefit from auditory training .

ELIGIBILITY:
Inclusion Criteria:

* Control group: (25) Children with normal peripheral hearing bilaterally their age is matched with the study group.
* Study group: three study groups, each study group has (25) children using, binaural Hearing aids, Cochlear implant and bimodal hearing with:
* Average IQ.
* No other congenital diseases affecting the speech progress.
* Using the hearing device for at least one year.
* Regular speech therapy sessions

Exclusion Criteria:

• Any other children not fulfilling the inclusion criteria or refuse to participate in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
speech process in the groups | 30 minutes after the test
  presence of the waves in the test traces

SECONDARY OUTCOMES:
best hearing amplification device | 30 minutes after the test
  best waves of the test traces

IPD SHARING:
Plan to Share IPD: No
The protocol

REFERENCES:
- [Result] Basoz Behmen M, Guler N, Kuru E, Bal N, Gedik Toker O. Speech auditory brainstem response in audiological practice: a systematic review. Eur Arch Otorhinolaryngol. 2023 May;280(5):2099-2118. doi: 10.1007/s00405-023-07830-3. Epub 2023 Jan 18. PMID 36651959
- [Result] Basu M, Krishnan A, Weber-Fox C. Brainstem correlates of temporal auditory processing in children with specific language impairment. Dev Sci. 2010 Jan 1;13(1):77-91. doi: 10.1111/j.1467-7687.2009.00849.x. PMID 20121865
- [Result] Walch C, Anderhuber W, Kole W, Berghold A. Bilateral sensorineural hearing disorders in children: etiology of deafness and evaluation of hearing tests. Int J Pediatr Otorhinolaryngol. 2000 Jun 9;53(1):31-8. doi: 10.1016/s0165-5876(00)00307-4. PMID 10862922
- [Result] Skoe E, Kraus N. Auditory brain stem response to complex sounds: a tutorial. Ear Hear. 2010 Jun;31(3):302-24. doi: 10.1097/AUD.0b013e3181cdb272. PMID 20084007
- [Result] Johnson KL, Nicol T, Zecker SG, Kraus N. Developmental plasticity in the human auditory brainstem. J Neurosci. 2008 Apr 9;28(15):4000-7. doi: 10.1523/JNEUROSCI.0012-08.2008. PMID 18400899
- [Result] Hood LJ. Auditory Neuropathy/Auditory Synaptopathy. Otolaryngol Clin North Am. 2021 Dec;54(6):1093-1100. doi: 10.1016/j.otc.2021.07.004. Epub 2021 Sep 15. PMID 34535280
- [Result] Davis A, Fortnum H, O'Donoghue G. Children who could benefit from a cochlear implant: a European estimate of projected numbers, cost and relevant characteristics. Int J Pediatr Otorhinolaryngol. 1995 Mar;31(2-3):221-33. doi: 10.1016/0165-5876(94)01115-e. PMID 7782180